CLINICAL TRIAL: NCT01557556
Title: Pexacerfont for Reduction of Stress-induced Tobacco Craving, Nicotine Reinforcement, and Brain Activation in Humans
Brief Title: Pexacerfont to Reduce Stress-induced Tobacco Craving
Status: Withdrawn | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912471; 12-DA-N471
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-12-16

CONDITIONS: Nicotine Dependence
Keywords: CRH Antagonist; Nicotine; Nicotine Dependence; Smoking; Stress
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Stressful situations often cause tobacco cravings. These cravings can make it very difficult for smokers who are trying to quit. Research has shown that craving may involve hormone pathways in the brain. The anti-anxiety drug pexacerfont acts on these hormone pathways. Researchers want to see if pexacerfont can act on the brain and lessen stress-related tobacco cravings in smokers who are trying to quit.

Objectives:

- To test the effects of pexacerfont on tobacco craving in smokers who want to quit smoking.

Eligibility:

- Smokers between 18 to 55 years of age who are trying to quit. (Participants must have smoked at least 10 cigarettes per day for at least 1 year.)

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will be assigned to take either pexacerfont or a placebo. They will take three pills every morning for the first 7 days, then one pill every morning for 23 days.
* At the first visit, participants will provide blood and urine samples. They will then be asked to prepare a 5-minute speech and give it to the study researchers. They will also be asked to do mental math problems for another 5 minutes. During these tests, blood pressure, heart rate, sweating, and skin temperature will be measured. Participants will fill out questionnaires about stress levels, tobacco cravings, and personal experiences.
* Participants will take the study pills for 30 days. Before the 2-week point, participants will be asked to try to quit smoking for 2 weeks.
* Participants will have four study visits. These visits will involve brain imaging scans and emotional stress tests. Tobacco cravings and other stress levels will be measured at each study. Blood and urine samples may be collected at these studies.
* Participants will have follow-up visits and phone calls for up to 6 months after the end of the study visits.

DETAILED DESCRIPTION:
Objective:

To evaluate pexacerfont, an orally available, brain-penetrant selective CRF1 antagonist, for its ability to modulate emotional and motivational processes in daily smokers who are seeking to quit smoking.

Study population:

We will collect evaluable data from up to 60 adult, greater than or equal to 10 cigarettes per day smokers who smoke their first cigarette within one hour of waking as reported on the Fagerstrom Test of Nicotine Dependence (FTND) and wish to quit smoking.

Design:

Participants will be randomly assigned to one of two groups to receive 30 days of oral pexacerfont (300 mg/day loading dose for 7 days, followed by 100 mg/day maintenance dose for 23 days) or matching placebo under double-blind conditions. On Day 15 and 16, subjects will have two days of testing to evaluate reactivity to stressful/neutral stimuli with and without the presence of smoking cues. Reactivity will be tested in terms of physiological parameters, subjective reports, nicotine reinforcemen, smoking resistance paradigms and functional Magnetic Resonance Imaging (fMRI) Blood Oxygen Level Dependent (BOLD) signal at rest and in response to stress/cue-related tasks. In addition, during the last 14 days of study drug administration, subjects will attempt to stop smoking. Daily assessments of smoking behavior will be obtained. Finally, on days 26 and 27, participants will again have two days of testing to evaluate reactivity to stressful/neutral stimuli. Reactivity will be tested in terms of physiological parameters, subjective reports, cue reactivity paradigms and functional Magnetic Resonance Imaging (fMRI) Blood Oxygen Level Dependent (BOLD) signal at rest and in response to stress/cue-related tasks.

Outcome measures:

Outcome measures in laboratory sessions will include nicotine reinforcement, latency to lapse in a smoking resistance paradigm, subjective ratings of stress, mood, and tobacco craving, autonomic responses (galvanic skin response, heart rate, and blood pressure), endocrine responses (salivary cortisol and salivary (alpha) amylase, a measure of endogenous adrenergic activity during stress), and fMRI BOLD signal at rest and in response to stress/cue-related tasks. Outcome measures during the quit attempt will include, change in consumption, number of lapses, and latency to lapse.

ELIGIBILITY:
* INCLUSION CRITERIA:

Daily smokers for at least one year; smoke at least 10 cigarettes per day; smoke first cigarette of day within one hour of waking as recorded on Fagerstrom Test of Nicotine Dependence (FTND).

Currently wish to quit smoking. Stage of Change (Prochaska and DiClemente, 1983) will be assessed for each participant and those who are in the contemplation and planning stages will be included in the study.

Urinary continine level greater than or equal to 100 ng/ml (NicAlert reading greater than or equal to 3) at screening.

Men and women, ages 18 to 55 years. Justification: Many cognitive processes change with age. In addition, the risk of difficult-to-detect medical abnormalities such as silent cerebral infarcts increases with age. As this study includes fMRI scanning, older individuals, defined as those over 55, will be excluded as these age-related abnormalities may affect quality of imaging data.

Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study drug, and agree to use an adequate method of contraception to avoid pregnancy from study entry to 6 months following the last dose of study drug. Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Adequate methods of contraception for sexually active women are having a male sexual partner(s) who is surgically sterilized prior to inclusion; having a sexual partner(s) who is/are exclusively female; using oral contraceptives (either combined or progestrogen only) with a single-barrier method of contraception consisting of spermicide and condom or diaphragm; using double-barrier contraception, specifically, a condom plus spermicide and a female diaphragm or cervical cap; or using an approved intrauterine device (IUD) with established efficacy.

Men, unless surgically sterilized (vasectomy with documentation of azoospermia), must agree to practice abstinence or use barrier contraception with spermacide (unless their partner has been surgically sterilized or is infertile), and not donate sperm, during drug administration and for a period of 6 months after the last dose of randomized treatment.

EXCLUSION CRITERIA:

Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Employees of BristolMyersSquibb (BMS) or immediate family of BMS employees.

People who are currently participating in another clinical study in which they are exposed to an investigational or non-investigational drug or device; people who have ever participated in a trial involving pexacerfont or closely related compounds.

People who are unable or unwilling to participate in an MR scan, including those who are left-handed, have metallic objects in the body (pacemaker, plates, clips, pins, rods, joints, pellets, cochlear implants, etc.), have pronounced claustrophobia, or who are physically incompatible with the machine dimensions.<TAB>

Women who are pregnant, breastfeeding, or planning to become pregnant within 6 months from the administration of last dose of study drug.

People with: Present Major Depressive Disorder, a past or present diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder; past or present diagnosis of dementia, or any other disorder which has led to a clinically significant cognitive impairment as assessed on screening evaluation by computerized SCID and clinical interview as well as the Wechsler Abbreviated Scale of Intelligence (WASI) vocabulary subtest with exclusion of participants with estimated full IQ less than 85.

People who currently use any illicit drugs or whose urine tests positive for illegal drugs at screening. People with a past history of dependence to drugs or alcohol, or who currently meet DSM-IV criteria for alcohol abuse or dependence or who consume more than 15 alcoholic drinks per week during the past month.

People with evidence of thyroid disease by medical history, on screening physical exam or

laboratory tests with TSH greater than 1.6 times upper limit of normal.

People with a current seizure disorder or a significant history (as judged by the investigators) of a seizure disorder, other significant neurological disorders (e.g., Parkinson s Disease, multiple sclerosis, stroke, neurodegenerative disease, cerebral palsy) or severe head trauma, or CNS tumor.

People with current renal or liver disease including abnormal liver function tests (LFT s): greater than or equal to 2.5 times upper limit of normal, Bilirubin 2 times upper limit of normal, or abnormal renal function: serum creatinine greater than or equal to 2mg/dL.

People with a history of diabetes mellitus type I and II or gastric bypass or reduction surgery. Justification: illnesses that change metabolism or the absorption from the GI tract, would interfere with drug metabolism or absorption).

People with cardiovascular abnormalities including diastolic BP greater than 105; systolic BP greater than 180; QTc greater than 475 msec.

People with hematologic abnormalities at screening: Platelets less than or equal to75,000/mm(3), hemoglobin less than or equal to 9g/dL, neutrophils, absolute less than or equal to 1000/mm(3).

People with HIV infection Justification: HIV can have CNS sequelae, thus introducing unnecessary variability into the data. Assessment tool(s): HIV salivary test.

People with difficulty swallowing capsules.

Current use or history of use in the last 3 months of psychiatric medications including but not limited to antidepressants, lithium, antipsychotics, anxiolytics, antiepileptics, opiates, or hypnotics.

Any change in a non-excluded medication in the past 3 months. If systemic intake of corticosteroids has occurred acutely within last 4 weeks or chronically within the last 6 months, one month should elapse since the last dose of systemic steroids before study drug initiation. (Topical hydrocortisone and inhaled corticosteroids are allowed).

Use of medications that are CYP3A4 inhibitors or inducers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02-24; Study Completion 2013-12-16

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)

REFERENCES:
- [Background] Bandettini PA, Wong EC. A hypercapnia-based normalization method for improved spatial localization of human brain activation with fMRI. NMR Biomed. 1997 Jun-Aug;10(4-5):197-203. doi: 10.1002/(sici)1099-1492(199706/08)10:4/53.0.co;2-s. PMID 9430348
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Binneman B, Feltner D, Kolluri S, Shi Y, Qiu R, Stiger T. A 6-week randomized, placebo-controlled trial of CP-316,311 (a selective CRH1 antagonist) in the treatment of major depression. Am J Psychiatry. 2008 May;165(5):617-20. doi: 10.1176/appi.ajp.2008.07071199. Epub 2008 Apr 15. PMID 18413705